CLINICAL TRIAL: NCT02811068
Title: An Observational Follow up Study of a Randomised Parallel Group Phase IV Study to Evaluate the Duration of the Immune Response to Vaccine and Non-vaccine HPV Types in UK Adolescent Females Who Received Either Cervarix or Gardasil Human Papillomavirus (HPV) Vaccines
Brief Title: Observational Follow up of Prior HPV Vaccinees
Acronym: HPVfollowup
Status: Completed | Type: Observational
Sponsor: Public Health England (Other Government)
Responsible Party: Sponsor
Other Study IDs: HPVfollowup
Record Dates: First submitted 2016-06-15; First posted 2016-06-23 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2018-08

CONDITIONS: Human Papillomavirus Virus
Keywords: HPV; vaccine; Human Papillomavirus Virus Vaccine
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — serology samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Venepuncture: Collection of single blood sample to assess antibody persistence over time
  Interventions: Other: venepuncture

INTERVENTIONS:
Other: venepuncture — single venepuncture

SUMMARY:
HPV vaccines have been included in the national immunisation schedule since 2008, firstly as the Cervarix vaccine which protects against two HPV types and in 2012 as the Gardasil vaccine which offers protection against a further two HPV types. This study will assess whether booster doses are indicated to protect females throughout their lifetime or if the vaccinations offered in early adolescence provide this by following up a cohort from a previous study where female adolescents were vaccinated 5-7 years ago.

DETAILED DESCRIPTION:
Since September 2008, Human Papillomavirus (HPV) vaccines have been offered as part of the UK national immunisation schedule to adolescent females, first as three doses of a bivalent vaccine (Cervarix) covering the two most common strains (HPV16 and 18). Subsequently a quadrivalent vaccine was given in 2012 (Gardasil) incorporating a further two HPV types (HPV6 and 11). Between 2009 and 2011, the National Vaccine Evaluation Consortium (NVEC) conducted a randomised, observer-blinded parallel group study to evaluate the immunogenicity of the two HPV vaccines in terms of humoral immune responses against vaccine and non-vaccine incorporated HPV genotypes. The investigators plan to approach the participants of the original study as part of a follow up study to assess the duration of the humoral immune response elicited to the HPV vaccines; specifically, comparing the breadth and magnitude of antibody responses against vaccine and non-vaccine incorporated genotypes 5.7-6.8years on from their first dose of vaccine.

Long-term follow up studies have been conducted up to 9.4 years post vaccination for example in a multicentre double-blinded trial evaluating the long term efficacy of the Cervarix vaccine, which demonstrated 95-100% sustained efficacy against incident infection and CIN1+/2+ lesions whilst antibody titres were above those seen with natural infection adding confidence to the long term efficacy of this vaccine . The quadrivalent vaccine has been evaluated in long term follow up studies for example in a continuation of the Future II study at 9 years post first dose, whereby ≥94% of samples were seropositive for types 6,11 and 16 and 60% for HPV18 according to a cut-off negative serostatus value decided on by a selection of naïve and seropositive sera. There was also minimal difference in titres compared to months 18 and 48, representing a stable plateau of seroprotective titres. There are only two studies that have examined the duration of antibody responses against non-vaccine genotypes beyond 12 months: one comparing antibody titers elicited by both HPV vaccines against HPV31 and HPV45 in 18-26 year old women 24 months post first dose and one describing HPV31 seropositivity in 18-25 year old women at 48 months. This study will therefore provide unique data for the age group that HPV vaccination is offered to in the UK, in terms of vaccine incorporated genotypes as there are a limited number of follow up studies evaluating the 12-15 year old age group, as well as assessing the duration of antibody responses against non-vaccine types which has been far less extensively studied in all age groups.

A minimum antibody titre that correlates with HPV vaccine efficacy has not been defined; that is, a so-called correlate of protection. For HPV16 and HPV18 this is, in part, due to the high levels of HPV antibody generated following vaccination and the lack of breakthrough infections in vaccine trials. For non-vaccine genotypes where efficacy is only partial, further information on the breadth, magnitude and duration of such antibody specificities is required before a correlate (or surrogate) of protection can be established .

There is evidence to suggest robust immunological memory from studies looking at booster doses of HPV vaccine, which could be introduced into the UK programme to ensure protection throughout a women's sexual lifetime. For instance, in a follow up study assessing the immunological response to a booster dose of Cervarix seven years following immunisation with a three dose schedule, a strong memory B cell response persists after vaccination, giving rise to significantly higher GMTs than observed following the first dose of the bivalent vaccine. A significant fold-increase in GMTs was also observed with a booster dose following two doses of the quadrivalent vaccine, though GMTs were higher following a bivalent booster.

This follow up study will begin to address the question of long term durability of HPV vaccine antibody responses afforded by the HPV vaccines in the target age group in the UK population and therefore whether changes need to be made to the current national schedule.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give written informed consent for participation.
* Females originally enrolled in the randomised parallel group study

Exclusion Criteria:

* Known bleeding diathesis (or any condition that may be associated with a prolonged bleeding time).
* Any other significant condition or circumstance which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: healthy volunteers who previously took part in a study of HPV vaccines
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
HPV immunogenicity | single timepoint per participant, over the duration of the study which is anticipated to be 12 months
  antibody titres elicited to HPV vaccine and non-vaccine types following vaccination with either Cervarix(R) or Gardasil(R) at 5-7 years post first immunisation and comparison between vaccines and over time

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Coates — Public Health England
Locations (2):
- United Kingdom (2):
  - Gloucestershire primary care, Gloucestershire, Gloucestershire
  - Hertfordshire primary care, Hertfordshire, Hertfordshire

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD